CLINICAL TRIAL: NCT00987909
Title: A Phase II Trial Assessing the Tolerability and Pharmacodynamic Effect of US SLIT Cat Hair in Subject With Cat Allergy and Investigating Efficacy Variables in an Environmental Exposure Chamber Model
Brief Title: Exposure Chamber Trial With Cat Immunotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Collaborators: Cetero Research, San Antonio (Network)
Responsible Party: Senior Director Global Clinical Development, ALK-Abelló A/S
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: US-C-01; Cetero Research - P2CR09001; Health Canada - 9427-A1556-24C
Record Dates: First submitted 2009-09-28; First posted 2009-10-01 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2010-08

CONDITIONS: Cat Allergy
Keywords: Cat; Allergy; Immunotherapy; Sublingual; Exposure chamber; Safety; Rhinoconjunctivitis
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Solution resembling the active solutions, but without allergen extract
  Interventions: Biological: Specific allergen immunotherapy (placebo)
- Cat hair allergen extract, dose group 1 (Experimental)
  Interventions: Biological: Specific allergen immunotherapy
- Cat hair allergen extract, dose group 2 (Experimental)
  Interventions: Biological: Specific allergen immunotherapy
- Cat hair allergen extract, dose group 3 (Experimental)
  Interventions: Biological: Specific allergen immunotherapy

INTERVENTIONS:
Biological: Specific allergen immunotherapy (placebo) — Drops for sublingual administration, 0 mcg (placebo), once daily administration for 16 weeks
  Arms: Placebo
Biological: Specific allergen immunotherapy — Drops for sublingual administration, 4.5 mcg Fel d1/day, once daily administration for 16 weeks.
  Arms: Cat hair allergen extract, dose group 1
Biological: Specific allergen immunotherapy — Drops for sublingual administration, 9.0 mcg Fel d1/day, once daily administration for 16 weeks
  Arms: Cat hair allergen extract, dose group 2
Biological: Specific allergen immunotherapy — Drops for sublingual administration, 18.0 mcg Fel d1/day, once daily administration for 16 weeks
  Arms: Cat hair allergen extract, dose group 3

SUMMARY:
The main purpose of this trial is to investigate if any of three different doses of cat hair immunotherapy is safe for treatment of cat allergic patients.

ELIGIBILITY:
Inclusion Criteria:

* A history of rhinoconjunctivitis on exposure to cats
* Positive Skin Prick Test response (wheal diameter at least 3 mm larger than the negative control
* Positive specific IgE against Fel d1 (at least IgE Class 2)
* Minimum qualifying rhinoconjunctivitis symptom score during EEC exposure at Visit 2

Exclusion Criteria:

* Uncontrolled asthma within the past 12 months, or asthma requiring regular use of inhaled corticosteroids
* FEV1 less than 80% of predicted
* Subjects who suffer from significant seasonal allergic rhinoconjunctivitis, and cannot complete the clinical trial outside the local pollen season, or who have significant allergy to other allergens (e.g. other animals or house dust mites) that cannot be avoided during the trial period
* Subjects who cannot tolerate baseline challenge in the Environmental Exposure Chamber
* History of anaphylaxis with cardio/respiratory symptoms
* A medical history of severe drug or food allergy with symptoms such as difficulty breathing, swelling of the face or a feeling of severe dizziness or increased heart rate
* Chronic urticaria
* History of severe cardiac disease
* Treatment with immunosuppressives, anti-IgE monoclonal antibodies, tricyclic antidepressants or MAOIs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events | During 16 weeks of treatment

SECONDARY OUTCOMES:
Rhinoconjunctivitis symptom score | After 0, 8, and 16 weeks of treatment
Overall rhinoconjunctivitis symptom score | After 0, 8, and 16 weeks of treatment
Acoustic Rhinometry | After 0, 8, and 16 weeks of treatment
Environmental Exposure Chamber Quality of Life | After 0, 8, and 16 weeks of treatment
Serum immunology | After 0, 8, and 16 weeks of treatment
Nasal secretion immunology | After 0 and 16 weeks of treatment
Safety lab testing (clinical chemistry, haematology, urinalysis) | After 0 and 16 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, CCFP, Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Cetero Research, Mississauga, Ontario, Canada